CLINICAL TRIAL: NCT02769819
Title: Identification of Morphological Characteristics to Predict Difficult Endotracheal Intubation Using a Flexible Fiberscope
Acronym: BFO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 16.051
Record Dates: First submitted 2016-05-10; First posted 2016-05-12 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Intubation; Difficult
Keywords: Flexible fiberscope

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intubation with a flexible fiberscope (Experimental): Following induction of general anesthesia and administration of a neuromuscular blocking agent, intubation will be performed using a flexible fiberscope.
  Interventions: Device: Flexible fiberscope

INTERVENTIONS:
Device: Flexible fiberscope — * Characteristics of patients will be assessed before induction of general anesthesia
  * Glottic visualization will be evaluated by direct laryngoscopy.
  * The endotracheal tube will be loaded onto the scope after silicon spray lubrication
  * Intubation will be performed with the flexible fiberscope with the patient in supine position with head and neck in neutral position
  * With the tip of the fiberscope in satisfactory position, the endotracheal tube will be advanced into the trachea. The scope will then be removed.
  * Accurate positioning of the endotracheal tube will be confirmed by capnography and lung auscultation.

SUMMARY:
This study is designed to identify patients' features predictive of difficult endotracheal intubation using a flexible fiberscope.

DETAILED DESCRIPTION:
Endotracheal intubation is an important act in the practice of anesthesiology. Direct laryngoscopy is the most commonly used technique to accomplish this task. Airway characteristics predicting difficult intubation with direct laryngoscopy are well defined. Physical findings, such as Mallampati classification or measurements of the thyromental distance, mouth opening, and neck extension have been validated to help anticipate difficult situations with the direct laryngoscope. When direct laryngoscopy is difficult, early conversion to an alternative technique reduces the risk of airway compromise and associated morbidity.

Many alternative intubation devices are now available, and part of the anesthesiologist's task is to select the alternative approach best suited to each patient's specific features. Despite its use for both elective and unexpectedly difficult intubation, predictive criteria for successful airway management with the flexible fiberscope have not been developed.

The purpose of this study is to identify patient morphometric or morphological characteristics, if any, that could predict difficult intubation when using the flexible fiberscope for perioperative tracheal intubation in an elective surgical population.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Patients undergoing elective surgery under general anesthesia, requiring endotracheal intubation

Exclusion Criteria:

* Induction planned without neuromuscular blocking agents
* Need for a rapid sequence induction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-09-12 (Actual); Study Completion 2017-09-12 (Actual)

PRIMARY OUTCOMES:
Morphologic and morphometric predictors of difficult intubation with the flexible fiberscope. | Patients will be followed from induction of anesthesia until the end of intubation, an average of 10 minutes
  This study will correlate patients' morphometric and morphologic characteristics with the number of attempts and time needed for intubation using a flexible fiberscope.

SECONDARY OUTCOMES:
Time to successful intubation | Patients will be followed from induction of anesthesia until the end of intubation, an average of 10 minutes
Number of attempts to successful intubation | Patients will be followed from induction of anesthesia until the end of intubation, an average of 10 minutes
Score on the Intubation Difficulty Scale | Patients will be followed from induction of anesthesia until the end of intubation, an average of 10 minutes
  To calculate the Intubation Difficulty Scale the following variables will be collected: number of attempts, number of operators, necessity to use an alternative intubation technique, glottic visualization and effort needed to obtain optimal view of the glottis, necessity of external laryngeal pressure and vocal cords position during intubation.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan R Williams, MD, PhD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Toure T, Williams SR, Kerouch M, Ruel M. Patient factors associated with difficult flexible bronchoscopic intubation under general anesthesia: a prospective observational study. Can J Anaesth. 2020 Jun;67(6):706-714. doi: 10.1007/s12630-020-01568-w. Epub 2020 Jan 17. PMID 31953669